CLINICAL TRIAL: NCT04256031
Title: Evaluation of the Effects of Smartphone Use on Posture, Pain, Function and Quality of Life in Young Adults
Brief Title: Effects of Smartphone Use on Posture, Pain, Function and QoL
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Sıla Yılmaz, Principal Investigator, Yeditepe University
Other Study IDs: YU1682
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Postural; Defect; Neck Pain, Posterior; Shoulder Pain; Quality of Life
Keywords: Smartphone addiction; Forward head posture; Rounded shoulder; Neck pain; Shoulder pain; Quality of life
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Internet Addiction Disorder | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Excessive Smartphone Use Group: Participants whose Smartphone Addiction Scale-Short Version scores are higher than 30
  Interventions: Other: Assessment
- Non-excessive Smartphone Use Group: Participants whose Smartphone Addiction Scale-Short Version scores are 30 or less
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The structured questionnaire, Visual Analogue Scale, Copenhagen Neck Functional Disability Scale, Shoulder Disability Questionnaire, World Health Organization Quality of Life Instrument-Short Form, and Smartphone Addiction Scale-Short Version will be applied to all participants respectively. Lastly, posture analysis will be performed to all participants by using the New York Posture Rating Chart.

SUMMARY:
The aim of the study is to determine the effects of the use of smartphone on the neck and shoulder posture, pain, and functions, and the quality of life in young adults. The sample of the study consists of university students. According to the scores they got from the Smartphone Addiction Scale-Short Version, all participants will be divided into two groups. The neck and shoulder posture, pain, and functions, and the quality of life will be compared between the two groups.

DETAILED DESCRIPTION:
The study will include 106 university students who are 18-25 years old. According to the scores they got from the Smartphone Addiction Scale-Short Version, all students will be divided into two groups as Excessive Smartphone Use Group and Non-excessive Smartphone Use Group, both consisting of 53 participants. Participants whose scores are higher than 30 will be included to the Excessive Smartphone Use Group, and whose scores are 30 or less will be included to the Non-excessive Smartphone Use Group. In the assessment of pain level, the Visual Analogue Scale will be used. Functional levels of the neck and shoulders will be evaluated with the Copenhagen Neck Functional Disability Scale and the Shoulder Disability Questionnaire. World Health Organization Quality of Life Instrument-Short Form will be utilized to assess the quality of life. Postural analyzes of the participants will be fulfilled with the New York Posture Rating Chart. All scores will be evaluated by comparing between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* To be willing and volunteer to participate in the study
* To be between 18 and 25 years old
* To have been using smartphone for more than 1 year

Exclusion Criteria:

* To have any health problem history or diagnosed pathology related with the neck or shoulder regions
* To have any history of trauma or surgery related to the neck or shoulder regions
* To have received any medical attention or treatment in the last six months because of a health problem related to neck or shoulder
* To have any diagnosed neurological problem

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample of the study will consist of university students.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-02-08 (Actual)

PRIMARY OUTCOMES:
Posture | 1 day (Instant single measure)
  Posture will be examined with New York Posture Rating Chart which is a quantitative approach to assess the alignment of various body parts from posterior and lateral. The total score calculated after the evaluation is at most 65, and at least 13. The low score indicates impairments in posture.
Pain level | 1 day (Instant single measure)
  In the assessment of the neck and shoulder pain levels the Visual Analogue Scale will be used. This scale is 10 cm long, and has two ends on a horizontal line. One of these two ends is called as "0", while one is named as "10". "0" point defines no pain, and "10" points describe the most severe pain.
Neck function | 1 day (Instant single measure)
  Functional level of the neck will be evaluated with the Copenhagen Neck Functional Disability Scale. It is a valid and reliable tool for self-assessment of cervical pain and related disabilities, developed by Jordan el al. in 1998. The minimum score of the scale is 0, while the maximum score is 30. Disability level increases as the total score increases.
Shoulder function | 1 day (Instant single measure)
  Functional level of the shoulder will be evaluated with the Shoulder Disability Questionnaire. It is a 16-items disability questionnaire related to shoulder pain. The result is calculated with a special formula, and evaluated out of 100. Disability level increases as the total score increases.
Quality of life level | 1 day (Instant single measure)
  World Health Organization Quality of Life Instrument-Short Form will be utilized to assess the quality of life of participants. This questionnaire has been developed by World Health Organization, and has been validated in 1999 by Eser et al. in Turkish population. The scale does not have a total score, each field of the scale is evaluated independently in itself and is scored out of 20 or 100 points. The higher the score shows the higher the quality of life level.
Smartphone addiction level | 1 day (Instant single measure)
  In determining the smartphone addiction levels of the participants, Smartphone Addiction Scale-Short Version will be utilized. It is a self-assessment tool questioning smartphone usage, constituted by Kwon et al in 2013. The validity and reliability study of its Turkish version was made by Noyan et al. in 2015. The cut-off score for Turkish population was detected both for male and female students in 2017 by Şata and Karip. The lowest score of the scale is 10, while the highest score is 60. As the score obtained from the scale increases, the severity of smartphone addiction increases.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmi Muammer, Professor, Study Chair — Yeditepe University, Department of Physiotherapy and Rehabilitation; Sıla Yılmaz, PT, Principal Investigator — Yeditepe University, Department of Physiotherapy and Rehabilitation
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akodu AK, Akinbo SR, Young QO. Correlation among smartphone addiction, craniovertebral angle, scapular dyskinesis, and selected anthropometric variables in physiotherapy undergraduates. J Taibah Univ Med Sci. 2018 Oct 5;13(6):528-534. doi: 10.1016/j.jtumed.2018.09.001. eCollection 2018 Dec. PMID 31435373